CLINICAL TRIAL: NCT06910488
Title: Daily Living Activities Mobile Application Program
Brief Title: The Effect of Daily Living Activities Mobile Application Developed for Individuals With Chronic Mental Disorder on Functionality
Acronym: RhMoGYA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, SENEM ONOL, Psychiatric nurse (Phd), Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Decision No: 22-2.1T/27
Record Dates: First submitted 2025-03-19; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Chronic Mental Disorders
Keywords: chronic mental disorders; mobile application; activities of daily living model; functionality; psychiatric nursing

STUDY DESIGN:
Intervention Model Description: In addition to routine rehabilitation services, activities of daily living mobile application programme was applied to the intervention group.
  The control group received routine rehabilitation services.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): In the study, an individual-specific rehabilitation programme consisting of diagnosis, planning and intervention stages was created for the patients included in the intervention group.
  In addition to routine rehabilitation services, the activities of daily living mobile application programme was applied to the intervention group in the form of face-to-face individual interviews, group training, use of RhMoGYA application by the patients for three months, and planning and follow-up of activities for the use of patients by the researcher.
  The interviews were planned within the scope of the Roper Activities of Daily Living Model for the development and follow-up of patients' activities of daily living.
  Interventions: Other: Daily Living Activities Mobile Application; Other: Individual interviews; Other: Group education; Other: Routine rehabilitation program
- Control group (Experimental): A routine rehabilitation program has been followed
  Interventions: Other: Routine rehabilitation program

INTERVENTIONS:
Other: Daily Living Activities Mobile Application — mobile application was used for three months
  Other Names: Experimental group
  Arms: Experimental group
Other: Individual interviews — The individual's daily living activities are assessed using forms and scales that evaluate disability, functional level, and the ability to perform skill-based activities.
  Factors affecting daily living activities, such as strengths and weaknesses, barriers, accessible healthcare services, and social support networks, are examined.
  The client's independent, semi-dependent, and dependent daily living activities are evaluated together.
  Implementation steps are created to achieve the identified goals. Barriers to achieving the goals and supporting factors are identified.
  Arms: Experimental group
Other: Group education — Information is provided about the symptoms of schizophrenia and bipolar disorder, their causes, and treatment.
  The early warning signs are explained, along with the importance of recognizing that they can lead to an emergency situation.
  The importance of prior planning for what to do in case of an emergency is discussed. As homework, the family is asked to make this plan together.
  Information is provided about the importance of daily living activities and what they entail.
  Information is provided about self-care skills, healthy nutrition, movement planning, good sleep hygiene, the importance of body temperature regulation, and elimination issues.
  Information is provided about communication skills. Information is given about what to pay attention to in order to establish effective communication.
  Arms: Experimental group
Other: Routine rehabilitation program — It includes psychiatric rehabilitation services that are part of the clinic's program.

SUMMARY:
The study was conducted to evaluate the functionality of a mobile application programme developed to help individuals with chronic mental disorders plan and implement their daily activities and its impact on activities of daily living.

The main questions it aims to answer are:

Does the activities of daily living mobile application programme improve participants' activities of daily living? Does the activities of daily living mobile application programme improve the activities of daily living? Does the activities of daily living mobile application programme improve participants' medication adherence?

DETAILED DESCRIPTION:
This study was conducted to evaluate the effect of a mobile application program developed to enable individuals with chronic mental disorders to plan and implement their daily activities on their functionality, daily activities, and medication adherence.

The study was designed as an experimental study with a control group, including pre-test, post-test, and follow-up measurements. A total of 64 patients with chronic mental disorders who met the inclusion criteria were included in the study, with 32 in the intervention group and 32 in the control group. Data were collected using the Introductory Information Form, the Social Functioning Assessment Scale (SFAS), the Lawton Instrumental Activities of Daily Living (IADL) Scale, and the Morisky Medication Adherence Scale (MMAS). Participants in the intervention group were administered the Activities of Daily Living-Based Mobile Application Programme developed in this study.

ELIGIBILITY:
Inclusion Criteria: - Individuals diagnosed with schizophrenia and bipolar disorder according to DSM-V

* Individuals aged between 18 and 65
* I've been in treatment for the last 3 months
* Can speak and understand Turkish
* Open to communication and co-operation
* Those who did not get 0 points from the phone usage step of the Lawton IADL (Lawton instrumental activities of daily living scale) data collection tool
* Android phone owner

Exclusion Criteria:

* Hearing, vision, speech and comprehension problems
* Individuals who did not attend the two scheduled sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Social Functioning Assessment Scale | Baseline and 5 months
  The evaluation range of the scale is 19 to 57 points. High score is interpreted as high level of functionality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Faculty of Medicine Hospital/ Department of Mental Health and Diseases, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: SAP, CSR
Time Frame: April 2025 - April 2026